CLINICAL TRIAL: NCT01471756
Title: Improving Complete Endoscopic Mucosal Resection (EMR) of Colorectal Neoplasia: A Randomized Prospective Comparison of Snares and Injectate in the Resection of Large Sessile Colonic Polyps
Brief Title: Improving Complete Endoscopic Mucosal Resection (EMR) of Colorectal Neoplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: US Endoscopy (Industry)
Responsible Party: Principal Investigator, Timothy Woodward, MD, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10-008104
Record Dates: First submitted 2011-09-29; First posted 2011-11-16 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms; Gastric Cancer
Keywords: sessile neoplasms; flat neoplasms; gastric cancer
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- iSnare with Gonak solution (Experimental)
  Interventions: Procedure: Standard of Care Procedure as described in ARM
- Snaremaster braided snare with Gonak solution (Experimental)
  Interventions: Procedure: Standard of Care Procedure as described in ARM
- iSnare with saline solution (Experimental)
  Interventions: Procedure: Standard of Care Procedure as described in ARM
- Snaremaster braided snare with saline solution (Experimental)
  Interventions: Procedure: Standard of Care Procedure as described in ARM

INTERVENTIONS:
Procedure: Standard of Care Procedure as described in ARM — Standard of Care Procedure as described in ARM

SUMMARY:
The investigators seek to compare two techniques of removing pre-cancerous lesions from the colon. The investigators also will compare two solutions used during the procedure to determine if either solution allows for an improved removal of the tumors.

DETAILED DESCRIPTION:
The primary aim of the study is to compare the efficacy, efficiency and safety of two types of snares used in Endoscopic Mucosal Resection (EMR), a combined needle and snare unit (ISnare, US Endoscopy) versus an oval braided snare with spiral wire (Snaremaster, Olympus). The secondary aim is to explore whether EMR efficacy and efficiency is depended upon the injection solution used, saline versus Gonak (a solution containing HPMC, saline, and epinephrine) for EMR.

ELIGIBILITY:
Inclusion Criteria:

* Sessile colorectal polyp
* laterally spreading lesions as defined by Paris Classification type II and > 1 cm or greater

Exclusion Criteria:

* Those with ulcerated depressed lesions (Paris type III) or biopsy proven invasive carcinoma
* Inflammatory bowel disease patients
* Coagulopathy ( INR> 1.5) that cannot be corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of Two Devices used in EMR | 1 year
  To explore the efficacy of two devices used in EMR (iSnare® system versus Snaremaster) as measured by the "Sydney Resection Quotient" (SRQ). SRQ is defined as "lesion size in mm divided by the number of pieces to resect" .

SECONDARY OUTCOMES:
Compare the Use of Two Injectates | 1 year
  To compare the use of two injectates (saline versus HPMC mixture) with respect to efficacy as measured by the aforementioned SRQ.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Woodward, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States